CLINICAL TRIAL: NCT00213720
Title: Place de l'Iode RadioActif Dans l'HyperThyroïdiE Sub-clinique (PIRHATES)/ Evaluation of the Interest of Subclinical Hyperthyroidism Treatment
Brief Title: Treatment of Subclinical Hyperthyroidism
Status: Terminated | Type: Observational
Why Stopped: recruitment difficulties
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 3463
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2020-09-29 (Actual); Status verified 2019-08

CONDITIONS: Subclinical Hyperthyroidism; Atrial Fibrillation
Keywords: Hyperthyroidism; atrial fibrillation; quality of life; radioiodine treatment
MeSH Terms: conditions — Atrial Fibrillation; Hyperthyroidism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum

SUMMARY:
Objective: To determine if the treatment of subclinical hyperthyroidism will reduce the rate of atrial fibrillation, the main complication of this condition.

DETAILED DESCRIPTION:
Randomized open-labelled multicentre study comparing radioiodine vs medical supervision without treatment

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 50 and greater
* Isolated decreased thyroid-stimulating hormone (TSH) with normal FT4 and FT3 levels

Exclusion Criteria:

* Iodide overload
* Non sinusal heart rhythm
* Severe heart disease

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients referred to tertiary hospitals for advice on thyroïd disease
Sampling Method: Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2005-08; Primary Completion 2019-11 (Actual); Study Completion 2020-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Goichot, MD, Principal Investigator — Hopitaux Universitaires de Strasbourg
Locations (21):
- France (21):
  - Patrick Roger, Bordeaux
  - Philippe Thiéblot, Clermont-Ferrand
  - Jean-Marcel Brun, Dijon
  - Jean-Louis Wemeau, Lille
  - Marie-Pierre Teissier, Limoges
  - Jacques Orgiazzi, Lyon
  - Bernard Conte-Delvox, Marseille
  - CH de Montbrison, Montbrison
  - Jacques Bringer, Montpellier
  - Marc Klein, Nancy
  - Michel Rodier, Nîmes
  - Laurence Leenhardt, Paris
  - Richard Marechaud, Poitiers
  - Brigitte Delemer, Reims
  - Claire Schvartz, Reims
  - Jean-Marc Kuhn, Rouen
  - Bruno Estour, Saint-Etienne
  - Centre Paul Strauss, Strasbourg
  - Hopitaux Universitaires de Strasbourg, Strasbourg
  - Philippe Caron, Toulouse
  - Pierre Lecomte, Tours